CLINICAL TRIAL: NCT04196010
Title: Dose-Finding (Phase 1) Study of Continuous Infusion Cladribine, Cytarabine and Mitoxantrone (CI-CLAM) for Adults With Relapsed/Refractory Acute Myeloid Leukemia or Other High-Grade Myeloid Neoplasms Treated at UW/SCCA
Brief Title: Continuous Infusion Chemotherapy (CI-CLAM) for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia or Other High-Grade Myeloid Neoplasms
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to unfavorable risk-benefit ratio of investigational regimen.
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1005551; NCI-2019-07696 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1005551 (Other: Fred Hutch/University of Washington Cancer Consortium); 10310 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2022-01

CONDITIONS: Myeloid Neoplasm; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
Keywords: Myeloid and Monocytic Leukemia; Other Hematopoietic
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute | interventions — Cladribine; Cytarabine; pegylated granulocyte colony-stimulating factor; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CI-CLAM, G-CSF) (Experimental): Patients receive CI-CLAM consisting of cladribine and cytarabine via CIV on days 1-2, 1-3, 1-4, 1-5, or 1-6 depending on dose level assignment, and mitoxantrone via CIV on days 1-2 or 1-3 depending on dose level assignment. G-CSF may be added at the discretion of the treating physician, as per standard of care. Patients that do not achieve a response of MRD-negative CR after the first cycle are eligible to receive a second cycle of CI-CLAM. Treatment continues for 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Biological: Recombinant Granulocyte Colony-Stimulating Factor; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Given subcutaneously
  Other Names: Recombinant Colony-Stimulating Factor 3; rhG-CSF; 143011-72-7
Drug: Mitoxantrone — Given IV
  Other Names: Dihydroxyanthracenedione; Mitozantrone

SUMMARY:
This phase I trial studies the side effects and best dose of a chemotherapy regimen given by continuous intravenous infusion (CI-CLAM), and to see how well it works in treating patients with acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory) or other high-grade myeloid neoplasms. Drugs used in CI-CLAM include cladribine, cytarabine and mitoxantrone, and work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Continuous intravenous infusion involves giving drugs over a time duration of equal to or more than 24 hours. Giving CLAM via continuous infusion may result in fewer side effects and have similar effectiveness when compared to giving CLAM over the shorter standard amount of time.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study.

Patients receive CI-CLAM consisting of cladribine and cytarabine via continuous intravenous infusion (CIV) on days 1-2, 1-3, 1-4, 1-5, or 1-6 depending on dose level assignment, and mitoxantrone via CIV on days 1-2 or 1-3 depending on dose level assignment. G-CSF may be added at the discretion of the treating physician, as per standard of care. Patients that do not achieve a response of minimal residual disease (MRD)-negative complete remission (CR) after the first cycle are eligible to receive a second cycle of CI-CLAM. Treatment continues for 2 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Initial presentation with > 10% myeloid blasts in peripheral blood or marrow and, after at least one course of induction treatment, now with > 5% blasts in peripheral blood or marrow, as assessed by morphology or multiparameter flow cytometry (MFC). Outside diagnostic material is acceptable if reviewed here. Patients may never have achieved an initial complete remission (< 5% blasts in marrow, absolute neutrophil count > 1,000 per microliter, platelet count > 100,000 per microliter) or may have relapsed from such a remission. Note that although "AML" is formally denoted by > 20% blasts and other high-grade myeloid neoplasm by 10-20% blasts, these two entities often have similar prognoses and respond similarly to therapy, with trials at University of Washington (UW)/Seattle Cancer Care Alliance (SCCA) as well as MD Anderson and various European cooperative groups not distinguishing between AML and other high grade myeloid neoplasms
* Treatment related mortality (TRM) score < 13.1
* Bilirubin < 2.0 mg/dl unless abnormalities thought due to organ infiltration by AML as suggested for example by white blood cell (WBC) > 25,000 and rising rapidly
* Creatinine < 2.0 mg/dl unless abnormalities thought due to organ infiltration by AML as suggested for example by WBC > 25,000 and rising rapidly
* Left ventricular ejection fraction > 45% by multigated acquisition scan (MUGA) scan or echocardiography, performed within 6 months prior to consent
* Off any active therapy for AML other than hydroxyurea for at least 1 week prior to study registration unless patient has rapidly progressive disease with resolution of all grade 2-4 non-hematologic toxicities. Patients with symptoms/signs of hyperleukocytosis or WBC > 100,000 and in whom there is a delay in scheduling a MUGA scan or other logistical delays can receive two doses of cytarabine (500 mg/m^2 each, but dosing is ultimately based on physician discretion)
* Men and women of childbearing potential must agree to use adequate contraception
* Not pregnant or lactating
* Not receiving other investigational agents
* Provision of informed written consent on study-specific consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 35 days from start of treatment (or 28 days only if a patient presents with an absolute blast count (white blood count x percent blasts) > 50,000 or one that is doubling every 3 days and is > 25,000)
  Will use the Bayesian Optimal Interval ("BOIN") design to select the MTDs for continuous infusion G-CSF, cladribine, cytarabine and mitoxantrone (CI GCLAM).

SECONDARY OUTCOMES:
Treatment responses | Up to 5 years post treatment
  Will assess treatment responses (e.g. complete response [CR] +/- minimal residual disease [MRD] , incomplete CR, morphologic leukemia free state, partial response, resistant disease).
Incidence of adverse events | Up to 5 years post treatment
  Will use the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for toxicity and adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Beth Percival, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT04196010/ICF_001.pdf